CLINICAL TRIAL: NCT03453671
Title: Strategies to Enhance the Experience of Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-0474
Record Dates: First submitted 2017-12-06; First posted 2018-03-05 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness; Osteogenesis, Distraction; Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will know their own condition (strategy) but not what the other conditions are. The primary investigator will be blind to participants' assignment to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (Experimental): Participants will use the strategy of mindfulness, i.e., present moment awareness with nonjudgment and acceptance, while exercising.
  Interventions: Behavioral: Mindfulness
- Distraction (Experimental): Participants will use the strategy of distraction, i.e., directing their attention to something other than exercise (specifically a podcast) while exercising.
  Interventions: Behavioral: Distraction
- Self-Monitoring (Active Comparator): Participants will monitor their internal experience while exercising, without distraction and without being taught mindfulness skills of nonjudgment and acceptance.
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Mindfulness — Participants will use mindfulness techniques while exercising
  Arms: Mindfulness
Behavioral: Distraction — Participants will distract themselves while exercising
  Arms: Distraction
Behavioral: Self-monitoring — Participants will use associative attentional focus while exercising
  Arms: Self-Monitoring

SUMMARY:
This study aims to test the effect of three cognitive strategies to affect individuals' subjective experience of cardiovascular exercise. Participants will be randomly assigned to one of three strategies to use while exercising, both during an in-person session and self-directed two week exercise period.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 40.
2. Insufficiently physically active for the past 6-months (i.e., does not meet American College of Sports Medicine [ACSM] guideline for cardiorespiratory exercise). The ACSM guidelines state that all healthy adults should engage in a minimum of 150 minutes per week of moderate intensity cardiorespiratory exercise, or 75 minutes per week of vigorous intensity exercise, or an equivalent combination of the two). On the eligibility screen assessment, we will define moderate and vigorous intensity exercise. Then we will ask individuals to report how many minutes of moderate and vigorous intensity exercise they engage in per week. We will use the ACSM's rule of thumb that 1 minute of moderate intensity exercise is equivalent to 2 minutes of vigorous intensity exercise. This will help to ensure that prospective participants who exercise for less than 150 minutes per week are not actually meeting the ACSM guidelines for cardiorespiratory fitness by engaging in vigorous intensity exercise. Thus, if total minutes of moderate intensity exercise and total minutes of vigorous intensity exercise (multiplied by 2) per week is equal to or greater than 150, callers will not be eligible for study inclusion.
3. Physically capable of safely engaging in moderate-intensity physical activity (PA)
4. Able and willing to access the Internet daily for two weeks
5. Willing to accept random assignment.
6. Have a smartphone or other mobile device (e.g., iPod Touch) that can play media (important if participants are assigned to the distraction condition)
7. Willing to engage in an exercise intervention specifically involving walking, jogging, running, or hiking (not other types of exercise)

Exclusion Criteria:

1. Are diabetic or receiving treatment for a metabolic disorder
2. Are currently pregnant
3. Are currently on antipsychotic medications
4. Have a history of cardiac or respiratory disease
5. Are receiving treatment for a heart condition or high blood pressure
6. Experience chest pains during and/or not during physical activity
7. Have a muscle, bone, or joint problem or injury that limit movement, make exercise painful, or could be made worse by exercising
8. Have a close family history of an adverse cardiac event before the age of 50.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals of all gender identities may participate in this study
Enrollment: 78 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Affective valence | 30 minutes
  Affective valence during a 30-minute exercise bout
Felt arousal | 30 minutes
  Felt arousal during a 30-minute exercise bout
Perceived Exertion (RPE) | 30 minutes
  Rating of Perceived Exertion during a 30-minute exercise bout
Minutes of exercise | 2-weeks following initial visit
  Minutes exercised during 2-week at-home intervention
Affect and perceived exertion: longitudinal | 2-weeks following initial visit
  Rated affect and perceived exertion during 2-week at-home intervention

SECONDARY OUTCOMES:
Theory of Planned Behavior: attitudes | Baseline to 2-week follow-up
  attitudes about exercise behavior
Theory of Planned Behavior: norms | Baseline to 2-week follow-up
  subjective norms regarding exercise behavior
Theory of Planned Behavior: self-efficacy | Baseline to 2-week follow-up
  self-efficacy for exercise
Theory of Planned Behavior Constructs | Baseline to 2-week follow-up
  intentions to engage in future exercise behavior
Distress tolerance | Baseline to 2-week follow-up
  Rated ability to tolerate distress
Defusion skills | Baseline to 2-week follow-up
  rated ability to "defuse"

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovation and Creativity (CINC), Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided